CLINICAL TRIAL: NCT00843375
Title: Evaluation of Stool Based Markers for the Early Detection of Colorectal Cancers and Adenomas
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Early Detection Research Network (Network); Clinical Genomics Pathology (Industry); VolitionRx (Unknown); Department of Health and Human Services (U.S. Federal Agency); Great Lakes New England Clinical Validation Center (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UMCC 2018.126 GLNE 007; U01CA086400 (NIH); HUM00149961 (Other: University of Michigan); UMCC 2018.126 (Other: University of Michigan); HUM00029506 (Other: University of Michigan); UMCC 2005.008 (Other: University of Michigan); HUM00161344 (Other: University of Michigan)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, up to 60 mls, will be obtained according to standard operating procedures. Subjects will collect stool samples per the schedule in the study calendar. Collection of Frozen Normal and Adenoma or Cancer Tissue: For individuals with large adenomas who are undergoing endoscopic resection, the fresh surgical sample will be obtained by the endoscopist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Higher risk, no neoplasia: Negative study colonoscopy and one or more of the following:
  * Subjects with a personal history of adenomas (confirmed by pathology) with none present on qualifying colonoscopy
  * Subjects with a personal history of colorectal cancer (CRC) (longer than 3 years ago because of exclusion criteria of cancer within last 3 years) with none present at time of qualifying colonoscopy
  * Any family history of CRC (1st degree relative)
  * Current positive screening stool test for blood, for DNA or for both within 12 months with no follow up intervention
- Adenoma: Pathologically confirmed adenomas, both non-advanced adenoma and advanced. Advanced adenoma includes any of the following:
  * Sessile serrated adenoma
  * Tubulovillous adenoma
  * Villous adenoma
  * Sessile serrated polyp/adenoma
  * Traditional serrated adenoma
  * Any adenoma ≥1 cm
- Colorectal adenocarcinoma: Pathologically confirmed colorectal cancer either present at time of stool collection or discovered during colonoscopy
- Average risk, no neoplasia: No neoplasia found at colonoscopy and:
  * No prior history of adenomas or sessile serrated adenomas
  * No prior history of CRC
  * No first degree family history of CRC
  * Negative colorectal cancer screening test (if performed) for blood, for DNA or for both within 12 months.

SUMMARY:
Colon cancer is the second most common cancer in men and women. It is a disease that can be prevented if it is found early. Colonoscopy is still the best screening tool for colon cancer and the polyps that turn into colon cancer. However, due to a variety of factors, including affordability, time, and age, not all patients are able to be screened. Researchers are working on other options for early detection that are as accurate as colonoscopy.

The purpose of this study if to determine if stool or blood can be used to detect colon cancers as early or earlier than colonoscopy. The researchers plan to use these samples to learn about specific proteins (also known as biomarkers) that may indicate colon polyps, colon cancer or an increased risk of developing colon cancer. In order to learn more about preventing and detecting colon and rectal cancer, we are collecting samples from subjects with cancer, adenomas, and colonoscopies who may be at risk for polyps.

DETAILED DESCRIPTION:
In recognition of the fact that novel potential biomarkers are continually being identified and will need to be validated in a rapid, efficient and scientifically rigorous manner, the NCI has made an enormous commitment to the development of a network that will facilitate biomarker development and validation in multiple organ sites. As part of the National Cancer Institute-funded Early Detection Research Network (EDRN), the Great Lakes-New England Clinical Epidemiological Center (GLNE CEC) proposes a research study that validates potential molecular markers ("biomarkers") for the detection of precancerous and cancerous conditions and cancer risk assessment. Although examples of such biomarkers are currently in clinical use (i.e. CEA, CA-125), there are limitations to all of them. Our consortium focuses on gastrointestinal neoplasia. The goals of this phase of the proposed research are:

1. Assessment of the utility of individual stool-based, serum-based and urine-based biomarkers for discriminating between patients with adenocarcinomas, patients with adenomas, patients without adenomas and normal subjects both at normal and high risk for developing colon cancer.
2. Construction of a panel of markers from those considered in Objective 1 to discriminate, under a number of assumptions concerning prevalence and cost of misclassification, between:

   1. Subjects with normal colons versus patients without adenomas, patients with adenomas and patients with cancers;
   2. Subjects with normal colons, patients without adenomas and patients with adenomas, versus subjects with cancers;
   3. Subjects with normal colons versus patients without and patients with adenomas versus patients with cancers.
3. Comparison of the characteristics of individual markers and panels as discriminators to those of the established current standard, fecal immunochemical test (FIT).
4. Continued support of a renewal of a bank of stool samples linked to serum, tissue, and clinical data from patients with colorectal cancer, adenomas and normal controls for validation of stool-based markers that may be developed in the future.

To build our collection, we propose to collect stool, FIT, serum, plasma, and tissue samples from 1200 new subjects. Each biomarker will be analyzed individually and considered as a potential panel marker to be used for future largescale screening longitudinal trials. (This protocol previously recruited an additional 682 subjects from January 2006 to June 2010.)

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent
* Able to physically tolerate removal of up to 60 ml of blood
* Adults at least 18 years old
* Willing to collect 1-2 stool samples and prepare a Fecal Immunochemical Test (FIT)
* Pregnant or nursing women who otherwise meet the eligibility criteria may participate
* Subjects with one of the following:

  * Colorectal adenocarcinoma-not treated and in colon at time of stool collection (CRC bin)
  * Adenoma-pathologically confirmed adenoma present in colon at time of stool collection (Adenoma Bin)
  * Higher Risk Non-neoplastic Bin

    * Subjects with a personal history of adenomas (confirmed by pathology) with none present on qualifying colonoscopy
    * Subjects with a personal history of CRC (longer than 3 years ago because of exclusion criteria of cancer within last 3 years) with none present at time of qualifying colonoscopy
    * Any family history of CRC (1st degree relative)
    * Current positive screening stool test for blood, for DNA or for both within 12 months with no follow-up intervention.
  * Average Risk, Non-neoplastic Bin

    * No history or current finding of any colorectal neoplasia including CRC, adenomas, sessile serrated adenomas and no family history of CRC.
    * Subjects who had CRC that was successfully treated at least three years ago may be considered eligible for the adenoma bin if their polyps are adenomas and there is no evidence of CRC, or for the higher risk non-neoplastic bin as noted above.
    * Subjects whose screening colonoscopy shows any of these types of polyps may be included in the non-neoplastic or the higher risk non-neoplastic bin if they meet the other criteria noted above.

      * Hyperplastic polyps
      * Benign mucosal polyps
      * Polypoid granulation tissue
      * Prolapsed mucosal polyps
      * Inflammatory polyp
      * Transitional mucosal polyp
      * Lipoma
      * Gangleoneuroma
      * Neuroma
      * Hamartomatous polyp

Exclusion Criteria:

* Cancer patients who have had any surgery, radiation, or chemotherapy for their current colorectal cancer prior to collecting the baseline samples
* History of or clinically active Inflammatory Bowel Disease
* Known HNPCC or FAP
* Inability to provide informed consent.
* Other active malignancy within 3 years of enrollment except any of the following:

  * Squamous cell carcinoma of the skin
  * Basal cell carcinoma of the skin
  * Carcinoma in situ of the cervix, Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery only. (Excluded if had pelvic radiation)
  * Stage Ia Grade 1 adenocarcinoma of the endometrium treated with surgery
* Patients on active chemotherapy or radiation treatment for any purpose
* Known HIV or chronic active viral hepatitis
* Women who are pregnant
* CT colonography (virtual colonoscopy) patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer and adenomas and scheduled for surgical or endoscopic resection or subjects scheduled for a colonoscopy will be recruited from collaborating consortium centers.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Retention: Samples with DNA | At 1 day of biospecimen collection
  Blood samples, up to 60 mls, will be obtained according to standard operating procedures. Subjects will collect stool samples per the schedule in the study calendar. Collection of Frozen Normal and Adenoma or Cancer Tissue: For individuals with large adenomas who are undergoing endoscopic resection, the fresh surgical sample will be obtained by the endoscopist.

CONTACTS AND LOCATIONS:
Overall Officials: Dean E Brenner, M.D., Principal Investigator — University of Michigan
Locations (13):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Carle Cancer Center, Urbana, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Langone Health, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Flinders Medical Center, Adelaide, South Australia, Australia
- St. Michael's Hospital, Toronto, Ontario, Canada